CLINICAL TRIAL: NCT04765072
Title: Expanding Rural Health Cancer Control Capacity: Focus on Cancer Survivorship
Brief Title: Expanding Rural Health Cancer Control Capacity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Debra Friedman (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Debra Friedman, Sponsor Investigator, Vanderbilt-Ingram Cancer Center
Organization: Vanderbilt-Ingram Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VICC PED 2019; 3P30CA068485-24S2 (NIH)
Record Dates: First submitted 2021-02-12; First posted 2021-02-21 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Survivorship care (Experimental): Participants in rural areas will receive a telehealth (providing health-related services through electronic communication technologies) survivorship care plan in combination with assistance from a patient navigator.
  Interventions: Behavioral: Survivorship Patient Navigation Intervention; Behavioral: Telehealth Survivorship Visit Intervention

INTERVENTIONS:
Behavioral: Survivorship Patient Navigation Intervention — Patient navigator assistance for navigating the healthcare system and locating and utilizing beneficial resources
Behavioral: Telehealth Survivorship Visit Intervention — Individualized survivorship care plan

SUMMARY:
Through this pilot study, investigators will test an innovative approach to implement survivorship care planning at three sites located in or adjacent to rural counties. The pilot data will inform a subsequent multi-site Hybrid Type 3 Implementation-Effectiveness study that will assess both implementation and clinical effectiveness outcomes.

DETAILED DESCRIPTION:
Study Aims:

* Pilot test the implementation of guideline-based survivorship care planning in a rural setting using patient navigation plus telehealth among underserved rural cancer survivors. Investigators will collect feasibility data on patient recruitment rates and the ability to measure clinical effectiveness outcomes using the electronic health record and patient reports (survivor adherence to recommended disease surveillance, health assessment and cancer prevention/early detection practices).
* Identify the facilitators and barriers to future larger scale implementation of guideline-based survivorship care planning in rural settings to optimize the implementation strategies. Through a mixed methods approach, investigators will address implementation research questions focused on "real world" implementation of the guideline-based intervention in rural areas, including barriers/facilitators and translation to other rural settings. This will allow us to optimize the implementation strategies that will be further evaluated in the future large-scale implementation trial

ELIGIBILITY:
Inclusion Criteria:

* Cancer patient at least 18 years of age at time of cancer therapy
* English-speaking with the ability to provide informed consent
* Received treatment for Stage 0 - III cancer with curative intent
* Completed cancer therapy within the previous 12 months (i.e., 12 months prior to consenting) and in complete remission

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Rate of improvement in adherence to survivorship plan (Survivorship Care Planning Experience Satisfaction Survey (1-5 Excellent - Poor) | Approximately 12 months
Measure effectiveness of Telehealth on survivorship care | Approximately 12 months
Estimate the facilitators to a future larger-scale implementation of guideline-based survivorship care planning in rural settings | Approximately 1 year
Estimate the barriers to a future larger-scale implementation of guideline-based survivorship care planning in rural settings | Approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Debra Friedman, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (4):
- United States (4):
  - Baptist Cancer Center- Golden Triangle Columbus, Columbus, Mississippi
  - Baptist Cancer Center - North Mississippi, Oxford, Mississippi
  - Baptist Cancer Center- Bartlett, Bartlett, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-23): https://cdn.clinicaltrials.gov/large-docs/72/NCT04765072/Prot_SAP_001.pdf
  • Informed Consent Form (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT04765072/ICF_000.pdf